CLINICAL TRIAL: NCT06361836
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Activity of Single Ascending Doses of SBT777101 in Subjects With Hidradenitis Suppurativa
Brief Title: Study of Single Doses of SBT777101 in Subjects With Hidradenitis Suppurativa
Acronym: Regulate-HS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sonoma Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SBT777101-02
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Hidradenitis Suppurativa
Keywords: regulatory T cells; CAR T; Treg; autologous; cell therapy; hidradenitis suppurativa; autoimmune disease; inflammatory disease
MeSH Terms: conditions — Hidradenitis Suppurativa; Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: Sequential escalating dose cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SBT777101 Dose Level 1 (Experimental): Low dose SBT777101
  Interventions: Biological: SBT777101
- SBT777101 Dose Level 2 (Experimental): Mid dose SBT777101
  Interventions: Biological: SBT777101
- SBT777101 Dose Level 3 (Experimental): High dose SBT777101
  Interventions: Biological: SBT777101

INTERVENTIONS:
Biological: SBT777101 — Experimental treatment

SUMMARY:
This study will test the safety and effects of SBT777101 when given as a single dose to subjects with hidradenitis suppurativa. Increasing dose levels will be given after the safety at lower dose levels is shown.

DETAILED DESCRIPTION:
The study evaluates the safety and effects of a novel regulatory CARTreg cell-based autoimmune and inflammatory disease therapy for the treatment of hidradenitis suppurativa. The therapy is an autologous (using the patient's own cells) Treg cell therapy that targets proteins in the inflamed, disease-associated tissue, with the aim to dampen inflammation and restore balance to the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≤50 kg/m2, inclusive
* Diagnosis of clinically active moderate-to-severe HS (Hurley Stage 2 or 3)
* Total abscess or inflammatory nodule (AN) count of ≥5, affecting at least 2 distinct anatomic regions, with at least 1 accessible AN of adequate size for biopsy (diameter > 1 cm)
* Total draining tunnel (dT) count of ≤20
* Documented history of inadequate response or intolerance to at least a 3-month course of 1 conventional systemic therapy (e.g., antibiotic) and 1 biologic drug (e.g., adalimumab or secukinumab)
* Doses of medications for HS must be stable for at least 5 weeks prior to study drug administration
* Must agree to use highly effective method of contraception for at least 1 year post SBT777101 administration

Exclusion Criteria:

* Major surgery within 12 weeks prior to screening or planned within 12 months after dosing
* History of or current inflammatory or other autoimmune disease
* Complex presentations of HS
* Skin disease other than HS that may confound clinical assessments or increase subject risk in the study
* Uncontrolled concomitant cardiovascular, nervous system, pulmonary, renal, hepatic, endocrine, or gastrointestinal disease
* Active current infection or history of recurrent infections
* Active or untreated latent tuberculosis
* Primary or secondary immunodeficiency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence, nature, and severity of adverse events [Safety and Tolerability] | Day of treatment to end of follow-up period (48 weeks)
Incidence and nature of Dose Limiting Toxicities [DLTs] | Day of treatment to end of DLT evaluation period (28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Arron, MD PhD, Study Director — Sonoma Biotherapeutics, Inc.
Locations (6):
- United States (6):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - SLUCare Academic Pavillion, St Louis, Missouri
  - Columbia University Irving Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No